CLINICAL TRIAL: NCT03327675
Title: High Precision Imaging of Prostate Specific Membrane Antigen for Personalized Treatment in Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S59428; 2016-003089-14 (EudraCT Number)
Record Dates: First submitted 2017-07-10; First posted 2017-10-31 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
Keywords: prostate-specific membrane antigen; Lymph Node Dissection; Prostatectomy; Positron-Emission Tomography
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; N,N'-bis(2-hydroxy-5-(ethylene-beta-carboxy)benzyl)ethylenediamine N,N'-diacetic acid; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA PET/MR (Experimental): Hybrid 68Ga-PSMA PET/MR scan
  Interventions: Other: 68Ga-PSMA (HBED-CC) PET

INTERVENTIONS:
Other: 68Ga-PSMA (HBED-CC) PET — 68Ga-PSMA PET/MR

SUMMARY:
This is an Investigator Initiated, non-commercial, single center, non-randomized, single arm, open label pilot study on 194 patients. The patients are affected by prostate cancer but in two different clinical settings. The first group is characterized by patients who are going to be operated of radical prostatectomy and they will undergo the study imaging preoperatively. The second group experiences biochemical relapse after primary treatment.

DETAILED DESCRIPTION:
Novel, sensitive tools, such as 68Ga-PSMA PET imaging, have great potential for very early disease detection and open the possibility of early curative local salvage treatment (with surgery, radiotherapy or a combination of both). This project will moreover provide important insights into the biodistribution and dosimetry of 68Ga-PSMA, opening possibilities of 90-Yttrium or 177-Lutetium-PSMA-based radionuclidetherapy of patients with metastatic PC in the future.

The study consists of 2 work units (WU):

Work-unit 1: Patients at high risk for nodal involvement prior to radical prostatectomy with extended lymph node dissection Work-unit 2: Biochemical recurrence after initial treatment with curative intent

ELIGIBILITY:
Inclusion criteria

Work-unit 1

* age < 75 years of age, with histologically proven invasive adenocarcinoma of the prostate
* a risk of equal or more than 5% of lymph node metastasis (intermediate to high risk disease), according to the Briganti nomogram (1)
* scheduled to undergo radical prostatectomy with extended lymph node dissection

Work-unit 2

* histologically proven diagnosis of prostate cancer
* biochemical relapse (two consecutive PSA≥0.2 ng/ml) of prostate cancer following radical local prostate treatment
* WHO performance state 0-1
* age > 18 years old

Exclusion criteria

Work-unit 1

* involvement of pelvic lymph nodes assessed by multi-parametric MRI
* evidence for bone metastasis assessed by bone scan (if PSA > 20 ng/ml)
* WHO performance status > 2
* previous pelvic irradiation or radical prostatectomy.
* other malignancy except adequately treated basal cell carcinoma of the skin diagnosed during the last 5 years
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Work-unit 2

* serum testosterone level <50ng/ml
* symptomatic metastases
* local relapse on MRI
* PSA rise while on active treatment with LHRH-agonist, LHRH-antagonist, Anti-androgen, Complete androgen blockade, Oestrogen-antioestrogen therapy
* previous treatment with cytotoxic agent for PCa
* treatment during the past month with products known to influence PSA levels (e.g. fluconazole, finasteride, corticosteroids,…)
* disorder precluding understanding of trial information or informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
68Ga-PSMA PET/MR imaging accuracy before radical prostatectomy + pelvic lymph node dissection [RP + PLND]. Work unit 1. 68Ga-PSMA PET/MR imaging accuracy in patients with biochemical recurrence after primary treatment. Work unit 2. | through study completion, an average of 2 year
  Assessment of the sensitivity, specificity, positive and negative predictive

SECONDARY OUTCOMES:
The correlation of tracer uptake to Gleason scores within the prostate tumor and within metastatic lymph nodes. Work unit 1. | through study completion, an average of 2 year
  Correlation between tracer uptake and pathology Gleason score
Comparison of diagnostic accuracy between 68Ga-PSMA PET, MR and combined 68Ga-PSMA PET/MR. Work unit 2. | through study completion, an average of 2 year
  Assessment of the sensitivity, specificity, positive and negative predictive value
The evaluation of change in patient management based on imaging results of 68Ga-PSMA PET/MR in patients with biochemical recurrence. Work unit 2. | through study completion, an average of 2 year
  Proportion of patients with treatments different from follow-up after the evaluation of 68Ga-PSMA PET/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Karolien Goffin, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

REFERENCES:
- [Derived] Draulans C, De Roover R, van der Heide UA, Kerkmeijer L, Smeenk RJ, Pos F, Vogel WV, Nagarajah J, Janssen M, Isebaert S, Maes F, Mai C, Oyen R, Joniau S, Kunze-Busch M, Goffin K, Haustermans K. Optimal 68Ga-PSMA and 18F-PSMA PET window levelling for gross tumour volume delineation in primary prostate cancer. Eur J Nucl Med Mol Imaging. 2021 Apr;48(4):1211-1218. doi: 10.1007/s00259-020-05059-4. Epub 2020 Oct 6. PMID 33025093